CLINICAL TRIAL: NCT06993116
Title: A Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-4712 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of SHR-4712 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4712-101
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-4712 Group (Experimental)
  Interventions: Drug: SHR-4712 Injection

INTERVENTIONS:
Drug: SHR-4712 Injection — SHR-4712 injection.

SUMMARY:
This is a Phase 1, open label, first-in-human study to evaluate safety, tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD), immunogenicity and anti-tumor activity of SHR-4712 in patients with advanced solid tumors. Patients will treat with SHR-4712 until unacceptable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates in this study and signs the informed consent form.
2. The subject is aged between 18 and 75 years old (inclusive), regardless of gender.
3. The subject must provide tumor tissue samples for biomarker testing.
4. The subject's ECOG performance status is 0 or 1.
5. The expected survival time is ≥ 12 weeks.
6. The subject has at least one measurable lesion that meets the requirements of RECIST v1.1.
7. Laboratory test results confirm that the subject has sufficient functions of vital organs.
8. Female subjects of child-bearing potential must not be breastfeeding, have no possibility of pregnancy, and agree to comply with relevant contraceptive requirements.

Exclusion Criteria:

1. The subject has a history of or currently has meningeal metastases, or has symptomatic and active central nervous system metastases.
2. The subject has spinal cord compression that has not been radically treated by surgery and/or radiotherapy.
3. The subject has uncontrollable tumor-related pain as judged by the investigator.
4. The subject has clinically symptomatic moderate or severe ascites, uncontrollable pleural effusion or pericardial effusion of moderate amount or more.
5. The subject has received systemic immunosuppressive treatment within 14 days before the first study drug administration.
6. The subject has active autoimmune diseases or a history of autoimmune diseases with a possibility of recurrence.
7. The subject has severe cardiovascular and cerebrovascular diseases.
8. The subject has other uncontrolled concomitant diseases before the first drug administration.
9. The subject has a history of severe allergic reactions to the test drug and its main formulation components.
10. The subject has a history of immunodeficiency, including positive HIV serological test results, and other acquired or congenital immunodeficiency diseases.
11. The subject has had a severe infection within 4 weeks before the first drug administration.
12. The subject has a history of active pulmonary tuberculosis infection within 1 year before enrollment as found through medical history or CT examination, or has a history of active pulmonary tuberculosis infection more than 1 year ago but has not received regular treatment.
13. The subject has other serious physical or mental diseases, known alcohol or drug dependence, abnormal laboratory test results, and other factors that may increase the risk of participating in the study or interfere with the study results, and any other situations that the investigator deems unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-06-09 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | First 21 days of treatment.
Adverse Events (AEs) | Approximately 24 months.

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) | Approximately 24 months.
Peak concentration (Cmax) | Approximately 24 months.
Trough concentration (Ctrough) | Approximately 24 months.
Area under the concentration-time curve from time zero to the last measurable time point (AUC0-t) | Approximately 24 months.
Area under the concentration-time curve from time zero to infinity (AUC0-∞) | Approximately 24 months.
Elimination half-life (t1/2) | Approximately 24 months.
Apparent clearance (CL/F) | Approximately 24 months.
Apparent volume of distribution (Vz/F) | Approximately 24 months.
Objective response rate (ORR) | Approximately 24 months.
Duration of objective tumor response (DoR) | Approximately 24 months.
Disease control rate (DCR) | Approximately 24 months.
Progression-free survival (PFS) | Approximately 24 months.
Overall survival (OS) | Approximately 24 months.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Undecided